CLINICAL TRIAL: NCT06897046
Title: Perioperative Study of Iparomlimab and Tuvonralimab in Resectable NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL-NSCLC-QIBA-1001
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); II-IIIB
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iparomlimab and Tuvonralimab combined chemotherapy neoadjuvant (Experimental): Neoadjuvant: Squamous Non-Small Cell Lung Cancer, Iparomlimab and Tuvonralimab 5 mg/kg Q3W (Day 1) + Paclitaxel（Albumin-bound ） 130 mg/m² Q3W (Day 1, Day 8) + Carboplatin (AUC=5) Q3W (Day 1) ; Non-Squamous Non-Small Cell Lung Cancer :Iparomlimab and Tuvonralimab 5 mg/kg Q3W (Day 1) + Pemetrexed 500 mg/m² Q3W (Day 1) + Carboplatin (AUC=5) Q3W (Day 1) Postoperative adjuvant therapy: Iparomlimab and Tuvonralimab combined chemotherapy or Iparomlimab and Tuvonralimab monotherapy or Other adjuvant treatment options
  Interventions: Drug: QL1706+Carboplatin+Paclitaxel（Albumin-bound ）/ Pemetrexed
- Iparomlimab and Tuvonralimab Neoadjuvant (Experimental): Neoadjuvant: Prior to surgery, participants receive 2-4 cycles Iparomlimab and Tuvonralimab, 5 mg/kg Q3W (Day 1). Postoperative adjuvant therapy: Iparomlimab and Tuvonralimab combined chemotherapy or Iparomlimab and Tuvonralimab monotherapy or Other adjuvant treatment options
  Interventions: Drug: QL1706

INTERVENTIONS:
Drug: QL1706 — PD-1/CTLA-4
  Arms: Iparomlimab and Tuvonralimab Neoadjuvant
Drug: QL1706+Carboplatin+Paclitaxel（Albumin-bound ）/ Pemetrexed — PD-1/CTLA4 combined chemotherapy drugs
  Arms: Iparomlimab and Tuvonralimab combined chemotherapy neoadjuvant

SUMMARY:
This project intends to study the efficacy and safety of Iparomlimab and Tuvonralimab with or without chemotherapyin the perioperative treatment of NSCLC

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntary Participation，willing to participate in this study and has signed the Informed Consent Form (ICF).

  2. Age, ≥18 years old, both male and female. 3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.

  4. Histologically or cytologically confirmed, treatment-naïve Stage II-IIIB (N2 only) non-small cell lung cancer (NSCLC) according to the 8th edition of the American Joint Committee on Cancer (AJCC). Only patients judged as T4 based on tumor size are allowed to be enrolled; other T4 conditions (e.g., invasion of the diaphragm, mediastinal involvement) are not permitted.

  5. The primary NSCLC is deemed resectable by multidisciplinary team (MDT) assessment, which must include a thoracic surgeon specializing in oncologic surgery.

  6. Ability to provide surgical or biopsy tumor tissue for biomarker analysis (e.g., genetic sequencing, PD-L1 testing). The following must be provided before enrollment: Formalin-fixed paraffin-embedded (FFPE) tissue block from within the past 3 months, or 5-10 unstained tissue slides, or 2 core biopsy specimens, along with the relevant pathology report. Fine-needle aspiration specimens are not acceptable.

  7. At least one measurable lesion according to RECIST v1.1 criteria, as determined by the investigator.

Exclusion Criteria:

* 1. Presence of confirmed EGFR or ALK positive mutations. 2. History of other malignancies within the past 5 years or concurrent malignancies, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell carcinoma of the skin, localized prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery.

  3. Previous treatment with immune checkpoint inhibitors (e.g., PD-1/PD-L1 agents), other drugs targeting T-cell receptors (e.g., CTLA-4), immune checkpoint agonist antibodies (e.g., anti-ICOS, CD40, CD137, GITR, OX40 antibodies), or anti-tumor immune cell therapy.

  4. History of Allogeneic Hematopoietic Stem Cell Transplantation or Solid Organ Transplantation: (except for corneal transplantation).

  5. Presence of congenital or acquired immunodeficiency (e.g., HIV infection). 6. History of severe allergic reactions to other monoclonal antibodies. 7. As determined by the investigator, any other factors that may affect study outcomes or lead to premature termination of the study, such as alcohol or drug abuse, other serious diseases (including psychiatric conditions) requiring concomitant treatment, significant laboratory abnormalities, or social or family factors that may impact patient safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-02-25 (Estimated); Study Completion 2027-05-25 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | 4 weeks after surgery
  pCR rate is defined as the percentage of patients, relative to the total of enrolled subjects,achieving complete histological regression with no available tumor cells

SECONDARY OUTCOMES:
Major Pathological Response Rate (MPR) | 4 weeks after surgery
  The MPR is defined as the percentage of subjects who underwent lung cancer resection with ≤10% residual viable tumor cells in the postoperative tumor bed (regardless of the presence or absence of residual viable tumor cells in the lymph nodes).
Objective Response Rate (ORR) | After completion of neoadjuvant therapy, before surgery
  The proportion of subjects who received neoadjuvant therapy and had at least one post-baseline imaging assessment, achieving a best response of complete response (CR) or partial response (PR) on preoperative imaging. For subjects who did not undergo surgical resection, the results from the first planned post-baseline imaging assessment were used for evaluation; confirmation of the best response was not required
R0 Resection Rate | 2 weeks after surgery
  The percentage of subjects who underwent resection and achieved complete resection (R0) among all subjects who received lung cancer surgery.
2-Year Event-Free Survival Rate (EFS) | up to 2 years
  Defined as the time from the date of first study treatment administration to the date of occurrence of any of the following events: disease progression or deterioration leading to inability to undergo surgery, attempted surgery but abandoned due to unresectable tumor or disease deterioration, postoperative disease progression or recurrence (RECIST 1.1), disease progression or recurrence without surgery, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Shugeng Gao, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Jie Wang, MD, Principal Investigator — Shanxi Province Cancer Hospital
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union, Beijing, China